CLINICAL TRIAL: NCT03842475
Title: Who Will Benefit From Bariatric Surgery for Diabetes? Using Fat Distribution Measurement, Gut Hormone Profiles and Genetic Data to Predict Diabetes Remission
Brief Title: Who Will Benefit From Bariatric Surgery for Diabetes?
Status: Recruiting | Type: Observational
Sponsor: Imperial College London (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor
Other Study IDs: IRAS:231300
Record Dates: First submitted 2019-01-31; First posted 2019-02-15 (Actual); Last update posted 2023-04-19 (Actual); Status verified 2023-04

CONDITIONS: Diabetes Mellitus, Type 2; Obesity
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity | interventions — Gastric Bypass

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Surgical cohort: Patients with type 2 diabetes undergoing Roux-en-Y gastric bypass surgery
  Interventions: Procedure: Roux-en-Y gastric bypass (RYGB)
- Control: Healthy volunteers with normal body mass index

INTERVENTIONS:
Procedure: Roux-en-Y gastric bypass (RYGB) — Bariatric surgery
  Groups: Surgical cohort

SUMMARY:
A study investigating the influence of fat distribution, genetic susceptibility markers for type 2 diabetes (T2DM) and fat distribution, epigenetic and transcriptomic changes and gut hormone responses to a mixed meal on diabetes remission following bariatric surgery.

ELIGIBILITY:
Bariatric surgery group

Inclusion Criteria:

* Males and females planning to undergo RYGB
* 18-80 years
* Type 2 diabetes mellitus or prediabetes
* Stable weight for at least 3 months
* Obese (BMI ≥30kg/m2)
* Eligible for surgery on the National Health Service (NHS) under The National Institute for Health and Care Excellence (NICE) 2014 criteria

Exclusion Criteria:

* Current pregnancy
* Inability to give informed consent
* Type 1 diabetes
* Low fasting C-peptide
* Secondary diabetes or absence of β-cell function
* Unable to undergo DEXA, cirrhosis, ascites, or other condition that may modify body fat composition e.g. underlying malignancy
* Current smoker
* Participation in another (interventional) trial within the last 3 months
* Unable to understand English

Healthy volunteers

Inclusion criteria:

* Aged 18-80 years
* Male or female
* Body mass index 19 - 25 kg/m2
* Stable weight for at least three months

Exclusion criteria:

* Abnormal glucose tolerance and fasting glucose
* History of any medical, or other condition, or use of any medications, including over-the-counter products, which, in the opinion of the investigators, would either interfere with the study
* Without access at home to a telephone, or other factor likely to interfere with ability to participate reliably in the study
* Pregnancy or breastfeeding
* Unable to maintain adequate contraception for the duration of the study
* Donated blood during the preceding 3 months or intention to do so before the end of the study
* Current smoker
* Participation in another trial within the last 3 months
* Unable to understand English

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Up to 150 patients recruited to completion from Imperial Weight Centre. Up to 60 healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 210 (Estimated)
Dates: Start 2018-10-01 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2028-10-05 (Estimated)

PRIMARY OUTCOMES:
Diabetes remission (partial or complete) | 1 year
Diabetes remission (complete) | 1 year

SECONDARY OUTCOMES:
Waist circumference, waist/hip ratio (cm) | 1 year
Body mass index (kg/m2) | 1 year
Weight loss | 1 year
Change in visceral adipose tissue | 1 year
  Dual Energy Xray Absorptiometry measurement (DEXA)
Change in visceral adipose tissue | 1 year
  Magnetic resonance imaging (MRI) measurement
Change in ectopic fat | 1 year
  MRI measurement

OTHER OUTCOMES:
Change in epigenetic data in tissues. | 1 year
Changes in the transcriptome in tissues | 1 year
Changes in gut hormone profiles | 1 year
Histological scoring of specimens for Non-alcoholic fatty liver disease/Non-alcoholic steatohepatitis | 1 year
Changes in gut microbiome | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Tricia Tan, MB ChB, Principal Investigator — Imperial College London
Locations (1):
- Imperial College Healthcare NHS Trust, London, Greater London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kenkre JS, Ahmed AR, Purkayastha S, Malallah K, Bloom S, Blakemore AI, Prevost AT, Tan T. Who will benefit from bariatric surgery for diabetes? A protocol for an observational cohort study. BMJ Open. 2021 Feb 10;11(2):e042355. doi: 10.1136/bmjopen-2020-042355. PMID 33568372